CLINICAL TRIAL: NCT03108703
Title: Assessment of Quality of Life and Outcomes in Patients Treated With Stereotactic Body Radiation Therapy (SBRT) for Primary Renal Cell Carcinoma (RCC) - AQuOS-RCC
Brief Title: Assessment of QoL and Outcomes With SBRT for RCC
Acronym: AQuOS-RCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Juravinski Cancer Center (Other)
Responsible Party: Principal Investigator, William Chu, MD, MSc, FRCPC, Radiation Oncologist, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 052-2015
Record Dates: First submitted 2017-03-19; First posted 2017-04-11 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Renal Cell Carcinoma
Keywords: RCC; Stereotactic Body Radiotherapy; SBRT; Stereotactic Ablative Radiotherapy; SABR
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SBRT (Experimental): RCC patients
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — 35-40 Gy delivered in 5 fractions

SUMMARY:
Stereotactic body radiotherapy (SBRT) is an emerging radiotherapy technique that precisely delivers high doses of radiation to tumours. It has been investigated as definitive treatment for an increasing variety of primary tumours including lung, liver, prostate, and now renal cell carcinoma (RCC). The principal aims of this study are to prospectively assess quality of life (QoL) and oncologic outcomes in non-surgical patients who receive SBRT for the treatment of RCC.

DETAILED DESCRIPTION:
There is an evolving body of literature that shows high rates of tumour control and minimal associated toxicities with SBRT to treat RCC. However, the majority of published evidence is retrospective in nature, and there is a scarcity of data on the impact on quality of life and cost-effectiveness of kidney SBRT.

The principal aims of this multicentre study are to prospectively assess QoL and oncologic outcomes in non-surgical patients who receive SBRT for the treatment of primary renal cell carcinoma.

The study population will include 30 consecutive patients treated with kidney SBRT on a conventional linear accelerator (35-40 Gy in 5 fractions) at the Odette Cancer Centre, Sunnybrook Health Sciences Centre, University of Toronto (OCC) and the Juravinski Cancer Center, Hamilton Health Sciences Centre, McMaster University (JCC).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old
* Medically inoperable or patient who refuses surgery
* Histologic diagnosis of RCC where possible, or radiologic evidence of growth on surveillance
* Lesion ≥2.5cm or recurrent lesion following local ablative therapy
* Written informed consent
* Participants must be able to understand the English-language or with the aid of a translator

Exclusion Criteria:

* ECOG ≥3
* Prior abdominal radiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-06; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Patient Quality of Life | Up to 5 years after treatment
  To evaluate quality of life scores

SECONDARY OUTCOMES:
Cost-Effectiveness | Up to 5 years after completion of treatment
  To assess health utility scores and correlate with QoL
Oncologic Outcomes | Up to 5 years after completion of treatment
  To evaluate local control
Oncologic Outcomes | Up to 5 years after completion of treatment
  To evaluate progression-free survival
Oncologic Outcomes | Up to 5 years after completion of treatment
  To evaluate overall survival
Treatment-Related Toxicity | Up to 5 years after completion of treatment
  To report number of participants with treatment-related toxicities as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Odette Cancer Centre, Sunnybrook Health Science Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No